CLINICAL TRIAL: NCT04518644
Title: Managed Access Program to Provide Access to Nilotinib, for Patients With Imatinib-intolerant and/or Resistant Ph+ Chronic Myelogenous Leukemia (CML) in Chronic Phase or CML in Accelerated Phase
Brief Title: Nilotinib, for Patients With CML-CP or CML-AP
Status: No longer available | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107A2411
Record Dates: First submitted 2020-08-14; First posted 2020-08-19 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Chronic Myelogenous Leukemia (CML)
Keywords: Nilotinib; Imatinib-intolerant; Imatinib resistant; Philadelphia Chromosome positive; Ph+; Chronic Myelogenous Leukemia in Chronic Phase; CML-CP; Chronic Myelogenous Leukemia in Accelerated Phase; CML-AP
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — nilotinib

INTERVENTIONS:
Drug: Nilotinib — The recommended dosing of nilotinib is 400 mg orally twice daily

SUMMARY:
The purpose of this Cohort Treatment Plan is to allow access to Nilotinib for eligible patients diagnosed with imatinib-intolerant and/or resistant Philadelphia Chromosome positive (Ph+) Chronic Myelogenous Leukemia in Chronic Phase (CML-CP) or Chronic Myelogenous Leukemia in Accelerated Phase (CML-AP). The patient's Treating Physician should follow the suggested treatment guidelines and comply with all local health authority regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. One of the diagnoses listed below

   * Imatinib resistant Philadelphia chromosome positive CML in chronic phase and the presence of the following criteria:
   * < 15% blasts in peripheral blood or bone marrow
   * < 30% blasts plus promyelocytes in peripheral blood and bone marrow
   * < 20 % basophils in the peripheral blood
   * ≥ 100 x 10^9 / L (≥ 100,000/mm3) platelets
   * No evidence of extramedullary leukemic involvement, with the exception of liver or spleen
   * Imatinib resistant Philadelphia chromosome positive CML in accelerated phase defined as never in blast crisis before starting treatment with one or more of the following criteria present within 4 weeks prior to beginning treatment:
   * ≥ 15% but < 30% blasts in blood or bone marrow
   * ≥ 30% blasts plus promyelocytes in peripheral blood or bone marrow (providing that <30% blasts present in bone marrow)
   * peripheral basophils ≥ 20%
   * thrombocytopenia < 100 x 10^9 / L unrelated to therapy
   * WHO Performance status of 0, 1, or 2
   * Imatinib must be discontinued at least 5 days prior to beginning nilotinib therapy
   * Normal organ, electrolyte and marrow functions as described below:

Potassium ≥ LLN (lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of investigational medication Total calcium (corrected for serum albumin) ≥ LLN or correctable with supplements Magnesium ≥ LLN or corrected to within normal limits with supplements prior to the first dose of investigational medication AST and ALT ≤ 2.5 x ULN or ≤ 5.0 x ULN if considered due to tumor Alkaline phosphatase ≤ 2.5 x ULN unless considered due to tumor Serum bilirubin ≤ 1.5 x ULN Serum amylase and lipase ≤ 1.5 x ULN Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥50 ml/min (calculated creatinine clearance using Cockcroft formula is acceptable) Serum phosphorous ≥ LLN or corrected to within normal limits with supplements prior to the first dose of nilotinib medication Written patient informed consent must be obtained prior to start of treatment. If consent cannot be expressed in writing, it must be formally documented and witnessed, ideally via an independent trusted witness. An acceptable alternative (e.g., an assent form, or consent from a parent or guardian) should be signed for legally incompetent patients (e.g., children).

Exclusion Criteria:

1. History of hypersensitivity to any drugs or metabolites of similar chemical classes as nilotinib.
2. Previous treatment with any cytotoxic investigational drug ≤4 weeks prior to beginning nilotinib. At least 2 weeks must have elapsed since the last dose of hormonal therapy or any approved or investigational "targeted" kinase inhibitor agent with the exception of imatinib which must be discontinued at least 5 days prior to beginning therapy with nilotinib.
3. Impaired cardiac function, including any one of the following:

   Inability to determine the QT interval on ECG Complete left bundle branch block Long QT syndrome or family history of long QT syndrome History of or presence of significant ventricular or atrial tachyarrhythmias Clinically significant resting brachycardia (<50 beats per minute) QTc > 450 msec on baseline ECG (using the QTcF formula). If QTc >450 and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient rescreened for QTc Myocardial infarction within 12 months prior to starting nilotinib Other clinically significant heart disease (e.g. unstable angina, congestive heart failure or uncontrolled hypertension).
4. any medications that prolong the QT interval and CYP3A4 inhibitors if the treatment cannot Use of be either safely discontinued or switched to a different medication prior to starting treatment. Please see http://crediblemeds.org/index.php for a comprehensive list of agents that prolong the QT interval
5. Severe and/ or uncontrolled concurrent medical disease that in the opinion of the treating physicians could cause unacceptable safety risks or compromise compliance with the compassionate use treatment (e.g. impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of nilotinib, ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection, uncontrolled diabetes, )
6. Patients who have undergone major surgery ≤ 2 weeks prior to Visit 1 or who have not recovered from side effects of such surgery
7. Known Cytopathologically confirmed Central Nervous System infiltration.
8. Use of therapeutic warfarin.
9. Acute or chronic liver or renal disease considered unrelated to tumor.
10. Treatment with any hematopoietic colony-stimulating growth factors ≤ 1 week prior to starting Nilotinib. Erythropoietin is allowed.
11. Patient who has not recovered from side effects of prior chemotherapy, immunotherapy, other investigational drugs, wide field radiotherapy, or major surgery. Patient who has received imatinib < 5 days prior to starting nilotinib or has not recovered from side effects of therapy. Hydroxyurea is permitted during the first 28 days of treatment (up to 5 g/day) for a maximum of 7 days.
12. Patient with a history of another primary malignancy that is currently clinically significant or requires active intervention.
13. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test (> 5 mIU/mL).
14. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, including women whose career, lifestyle, or sexual orientation precludes intercourse with a male partner and women whose partners have been sterilized by vasectomy or other means, UNLESS they are using two birth control methods. The two methods can be a double barrier method or a barrier method plus a hormonal method.

Adequate barrier methods of contraception include: diaphragm, condom (by the partner), intrauterine device (copper or hormonal), sponge or spermicide. Hormonal contraceptives include any marketed contraceptive agent that includes an estrogen and/or a progestational agent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult